CLINICAL TRIAL: NCT04253067
Title: A Single-Blind, Randomized Study to Compare the Efficacy and Safety of Fractional Carbon Dioxide Laser Therapy Versus Sham for Treatment of Stress Urinary Incontinence Symptoms in Women
Brief Title: A Single-Blind, Randomized Study to Compare fCO2 Laser Therapy Versus Sham for Treatment of SUI in Women
Acronym: LaserSUI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided not to open study, following review of data collected in another study
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-LaserSUI
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Stress Urinary Incontinence; Urinary Incontinence
Keywords: Laser Therapy
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to active fCO2 laser therapy or sham. Study will be performed in a single-blind manner. (Participant and biostatistician)
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blind, participant and biostatistician will be blinded to treatment group. Subjects will be randomized 1:1 to active fCO2 laser treatment group or sham treatment group. Randomization will be performed using a table of random numbers. Randomization envelopes will be provided by the biostatistician and will be securely stored in a locked cabinet. The research coordinator(s) will be responsible for maintaining the confidentiality and security of the randomization envelopes. An enrollment and randomization log will be stored securely. The biostatistician will prepare more envelopes, if necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active fCO2 laser treatment (Active Comparator): Laser probe will be inserted into the vagina. The laser treatment is delivered at 6 points to the vaginal wall. Delivery begins at the most proximal and the wand is retracted by 1 cm and another row of laser treatment is delivered. The number of levels is determined by vaginal length.
  Interventions: Device: Active fCO2 laser treatment
- Sham fCO2 laser treatment (Sham Comparator): Laser probe will be inserted into the vagina. To prevent the delivery of laser energy, the laser will remain in standby mode during the visit. Keeping the laser in standby mode prevents laser exposure. The treatment will appear to be the same as the active treatment. The machine maintains a low humming noise while in standby mode.
  Interventions: Device: Sham fCO2 laser treatment

INTERVENTIONS:
Device: Active fCO2 laser treatment — The laser probe is inserted into the vagina. Laser treatment is delivered at 6 points at each level of the vaginal wall (12, 2, 4, 6, and 10 o'clock positions). Delivery begins at the most proximal and the probe is retracted by 1 cm and another row of laser treatments are delivered. The number of levels is determined by the patient's vaginal length.
  Arms: Active fCO2 laser treatment
Device: Sham fCO2 laser treatment — The laser probe is inserted into the vagina. The laser will remain in standby mode during the treatment preventing laser exposure. The treatment will appear to be the same as the active treatment with the probe starting at the most proximal and following the same 6 points of treatment delivery. The probe is retracted in the same manner and another row of treatment is simulated. The machine maintains a low humming noise while in standby mode. No active laser treatment is delivered.
  Arms: Sham fCO2 laser treatment

SUMMARY:
This is a prospective randomized sham-controlled study of patients undergoing vaginal treatment with a fractional carbon dioxide (fCO2) laser for stress urinary incontinence (SUI) symptoms. Eligible participants will be randomized (like a flip of a coin) to receive active or sham fCO2 laser treatments. Three treatments with the fCO2 laser or sham to the vagina will be performed, approximately four weeks apart.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is a common problem that affects 35-40% of women worldwide. SUI occurs when a woman experiences involuntary leakage of urine with physical activities such as exercise, coughing and sneezing that increases intra-abdominal pressure. Vaginal laser therapy offers a potential novel treatment for SUI, however there is limited scientific evidence to show benefits to treatment. A sham controlled study will further add to the literature and evidence to support or oppose the use of the fCO2 laser for SUI.

The purpose of this study is to compare active therapy to sham treatment to determine if a true benefit to treatment exists. Eligible participants will be randomized 1:1, to receive active or sham fCO2 laser treatments. Three treatments, active or sham, to the vagina will be performed approximately four weeks apart. The primary efficacy endpoint is four weeks after completing all treatments. Treatment durability and safety will be assessed eight weeks after the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age ≥18 years and ≤75 of age
3. Mild to moderate SUI defined by Stamey Grade 1 and 2
4. Positive bladder stress test at screening
5. Negative urinary tract infection (UTI) at the time of study enrollment. If a patient does have a UTI, they may be rescreened after treatment
6. No additional SUI therapy in the past 2 months such as pelvic floor physical therapy, medications, or participation in another SUI study
7. No prior history of midurethral sling or fascial sling for SUI
8. No prior history of urethral bulking procedure for SUI
9. No prior history of autologous muscle derived stem cell injection in the urethra
10. Must sign the informed consent form
11. Must be willing to comply with the study protocol

Exclusion Criteria:

1. Contraindications to fCO2 laser treatment, such as:

   1. previous pelvic mesh surgery
   2. current or previous genital cancers,
   3. radiation to the vaginal or colo-rectal tissue,
   4. currently pregnant or less than 3 months following pregnancy
   5. active infections (candidiasis, herpes genitalis, etc.)
   6. vaginal or cervical lesions noted on initial exam
2. Patients with undiagnosed vaginal bleeding not related to menses
3. Active vulvar or vaginal infection, including herpes
4. Current UTI, confirmed by positive urine culture and patient-reported UTI symptoms
5. Recurrent UTI defined as 3 UTIs in the past 6 months or 4 UTIs in the past 1 year
6. Pelvic or vaginal surgery within the past 9 months
7. Pelvic organ prolapse beyond the introitus
8. Patient possesses any other characteristics that, per the investigator's judgment, deems them unsuitable (i.e. may increase patient's risk, may affect the conduct of the study, etc.) for the treatment and/or study.
9. Participation in an investigational trial that used a study treatment, medication and/or biologic within 30 days or less prior to the date of the screening visit.

Deferral

Patients may be deferred and rescreened at a later date under the following conditions:

* Patients with active vulvar or vaginal infections may be rescreened after treatment
* Patients with an active UTI may be rescreened after treatment
* Patients with undiagnosed vaginal bleeding may be rescreened after complete work-up, treatment and resolution of vaginal bleeding
* Patients pregnant within the past 3 months
* Patients with recent vaginal or uterine surgery within the 9 months

Note: To preserve the scientific integrity of the study some inclusion and exclusion criteria are not listed. At the conclusion of the study all items will be posted.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of fCO2 laser therapy in women with mild to moderate SUI symptoms compared to sham by evaluating the responder rate. | 4 weeks after completing all treatments
  A patient is called a responder if there is a greater than or equal to 50% reduction from baseline in the number of subject-reported SUI episodes over 3 days on a voiding diary.

SECONDARY OUTCOMES:
To compare fCO2 laser therapy vs. sham in relation to the change in the total number of voids per day as measured by the 3-day voiding diary. | 8 weeks after the primary endpoint
  Change in the total number of subject-reported stress urinary incontinence (SUI) episodes over 3 days based on voiding diaries. Each void and urine leak will be recorded over a 3 day period. Patients will determine if each leak is a stress leak or urge leak. Patients will be given a 3 day diary to complete.
To compare fCO2 laser therapy vs. sham in relation to the change in subject-reported impression of SUI severity. | 8 weeks after the primary endpoint
  SUI severity as measured by the Patient Global Impression of Severity Scale (PGI-S). The subject will check the box that describes how their condition is now. Available options are 1= normal, 2 = mild, 3 = moderate, or 4 = severe. A higher score is equivalent to a worse outcome.
To compare fCO2 laser therapy vs. sham in relation to the change in subject-reported impression of SUI improvement. | 8 weeks after the primary endpoint
  SUI improvement as measured by the Patient Global Impression of Improvement Scale (PGI-I). The subject will select one of the following options, (very much better, much better, a little better, no change, a little worse, much worse, very much worse) to describe their SUI symptoms now versus prior to study treatment.
To compare fCO2 laser therapy vs. sham in relation to the change in subject-reported urogenital distress. | 8 weeks after the primary endpoint
  Change in urogenital distress as measured by the Urinary Distress Inventory questionnaire (UDI-6). The UDI-6 is a six point questionnaire, each question is scored as follows: 0 = no, 1 = not at all, 2 = somewhat, 3 = moderately, 4 = quite a bit. Scores are totaled and divided by 6, then multiplied by 25 to calculate the raw score. Higher scores = higher disability.
To compare fCO2 laser therapy vs. sham in relation to the change in subject-reported impact of urinary incontinence on daily life as measured by the Incontinence Impact Questionnaire (IIQ-7). | 8 weeks after the primary endpoint
  Impact of urinary incontinence on daily life as measured by the Incontinence Impact Questionnaire (IIQ-7). The IIQ-7 assesses how a subject's problem effects activities, relationships, and feelings. It is a 7 point questionnaire. Each answer is scored as: 0=not at all, 1=slightly, 2=moderately, 3=greatly. The higher the score the more effected they are by their condition.
To compare fCO2 laser therapy vs. sham in relation to the change in subject-reported impact of urinary incontinence on daily life as measured by the Incontinence Quality of Life Questionnaire (I-QOL) | 8 weeks after the primary endpoint
  The impact on urinary incontinence as measured by the Incontinence Quality of Life questionnaire (I-QOL). The I-QOL is a quality of life measure specific to persons with urinary incontinence. The survey consists of 22 incontinent-specific quality of life items, all having the following five-point ordinal response; 1=extremely, 2=quite a lot, 3=moderately, 4=a little, 5=not at all. The summed total score is transformed to a 0-100 scale ranging from 0 (poor quality of life) to 100 (maximum quality of life).
To compare fCO2 laser therapy vs. sham in relation to the change in subject-reported fecal incontinence. | 8 weeks after the primary endpoint
  Change in fecal incontinence as measured by the Cleveland clinic incontinence score (Wexner). Incontinence of stool may occur with or without urinary leakage. On the Cleveland clinic incontinence score the type of incontinence of stool (solid, liquid, gas, wears pad, lifestyle altered) are reported by the subject. Each question is measured as 0=never, 1=rarely, 2=sometimes, 4=usually, 5=always. The higher the score the more severe the condition.
To compare fCO2 laser therapy vs. sham in relation to the change in subject-reported sexual function. | 8 weeks after the primary endpoint
  Change in sexual function as measured by the Female Sexual Function Index Questionnaire (FSFI). The FSFI is a 19 question survey. A lower score is equivalent to a higher degree of sexual function. Scores range from 0 to 95.
To compare fCO2 laser therapy vs. sham in relation to the change in subject-reported pain and discomfort. | 8 weeks after the primary endpoint
  Change in pain and discomfort as measured by the Visual Analog Scale (VAS). The VAS is a validated questionnaire that assesses pain on a scale from 0=no pain to 10=Worst possible pain. A higher score is equivalent to a worse outcome.
Durability to determine whether subjects in the fCO2 laser therapy group continue to have a higher responder rate than the sham group. | 8 weeks after the primary endpoint.
  A patient is called a responder if there is a greater than or equal to 50% reduction from baseline in the number of subject-reported SUI episodes over 3 days on a voiding diary. Change in the total number of subject-reported stress urinary incontinence (SUI) episodes over 3 days based on voiding diaries. Each void and urine leak will be recorded over a 3 day period. Patients will determine if each leak is a stress leak or urge leak. Patients will be given a 3 day diary to complete.
Determine the safety of fCO2 laser therapy compared to sham. | 8 weeks after the primary endpoint.
  Safety of the fCO2 laser therapy compared to sham will be assessed in relation to the incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, Principal Investigator — Beaumont Hospital-Royal Oak
Locations (1):
- Beaumont Hospital-Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601